CLINICAL TRIAL: NCT02216461
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Inhaled Doses (7.5 to 60 mg Daily for 12 Days) of BIBW 2948 BS Inhalation Powder, Hard Capsule for HandiHaler® in Healthy Male Volunteers (Randomised, Double-blind Placebo-controlled Within Dose Groups)
Brief Title: Safety, Tolerability and Pharmacokinetics of BIBW 2948 BS for HandiHaler® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1219.3
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Inhalation

ARMS (4):
- Low dose of BIBW 2948 BS (Experimental)
  Interventions: Drug: Low dose of BIBW 2948 BS for oral inhalation
- Medium dose of BIBW 2948 BS (Experimental)
  Interventions: Drug: Medium dose of BIBW 2948 BS for oral inhalation
- High dose of BIBW 2948 BS (Experimental)
  Interventions: Drug: High dose of BIBW 2948 BS for oral inhalation
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose of BIBW 2948 BS for oral inhalation
  Arms: Low dose of BIBW 2948 BS
Drug: Medium dose of BIBW 2948 BS for oral inhalation
  Arms: Medium dose of BIBW 2948 BS
Drug: High dose of BIBW 2948 BS for oral inhalation
  Arms: High dose of BIBW 2948 BS
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability, and pharmacokinetics of BIBW 2948 BS after repeated dosing

ELIGIBILITY:
Inclusion Criteria:

* Healthy males based on a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥21 and Age ≤ 50 years
* BMI (Body Mass Index) ≥18.5 and BMI ≤ 29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation
* Subjects must be current smokers (<10 cigarettes or <3 cigars <3 pipes/day) with a smoking history >1 year

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which may have reasonably influenced the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-01; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant findings in vital signs | Up to day 20 after start of treatment
Number of patients with clinically significant findings in 12-lead electrocardiogram (ECG) | Up to day 20 after start of treatment
Number of patients with clinically significant findings in clinical laboratory tests | Up to day 20 after start of treatment
Number of patients with adverse events | Up to day 41
Assessment of tolerability by investigator on a 4-point scale | Up to day 20 after start of treatment

SECONDARY OUTCOMES:
Maximum concentration of the analyte BIBW in plasma at different time points (Cmax) | Pre-dose, up to 336 hours after start of treatment
Time from dosing to maximum measured concentration of the analyte in plasma at different time points (tmax) | Pre-dose, up to 336 hours after start of treatment
area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ (AUCτ,1) | Pre-dose, up to 336 hours after start of treatment
The percentage of the area under the concentration-time curve of the analyte in plasma over the time interval from 0 to infinity (AUC0-∞) that is obtained by extrapolation (%AUCtz-∞) | Pre-dose, up to 336 hours after start of treatment
Terminal rate constant of the analyte in plasma at different time points (λz) | Pre-dose, up to 336 hours after start of treatment
Terminal half-life of the analyte in plasma at different time points (t1/2) | Pre-dose, up to 336 hours after start of treatment
Mean residence time of the analyte in the body after one administration at different time points (MRTih) | Pre-dose, up to 336 hours after start of treatment
Apparent clearance of the analyte in plasma following extravascular administration at different time points (CL/F) | Pre-dose, up to 336 hours after start of treatment
Apparent volume of distribution during the terminal phase λz following an extravascular administration at different time points (Vz/F) | Pre-dose, up to 336 hours after start of treatment
Amount of analyte that is eliminated in urine from at different time points (Ae) | Pre-dose, up to 336 hours after start of treatment
Fraction of analyte eliminated in urine at different time points (fe) | Pre-dose, up to 336 hours after start of treatment
Renal clearance of the analyte at different time points (CLR) | Pre-dose, up to 336 hours after start of treatment
Minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | Pre-dose, up to 336 hours after start of treatment
Accumulation ratio of the analyte in plasma after multiple dose administration over a uniform dosing interval τ based on Cmax (RA,Cmax,10) | Pre-dose, up to 336 hours after start of treatment
Accumulation ratio of the analyte in plasma after multiple dose administration over a uniform dosing interval τ based on AUC0-τ (RA,AUC,10) | Pre-dose, up to 336 hours after start of treatment
Linearity index (AUCτ,ss / AUC0-∞) | Pre-dose, up to 336 hours after start of treatment
Changes from baseline in induced sputum analysis (amount of cells, mucin) | Pre-dose, 268 hours after start of treatment
area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Pre-dose, up to 336 hours after start of treatment
area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable concentration at tz (AUC0-tz) | Pre-dose, up to 336 hours after start of treatment